CLINICAL TRIAL: NCT00859638
Title: I Am Able: Population Based Rehabilitation in a Family Health Team
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Responsible Party: Dr. Julie Richardson, McMaster University
Organization: McMaster University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08-177; 2007-ORRAN-IIA-568
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Results first posted 2010-06-17 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Conditions; Arthritis; Diabetes; Hypertension; Chronic Pain
MeSH Terms: conditions — Chronic Disease; Arthritis; Diabetes Mellitus; Hypertension; Chronic Pain | interventions — Physical Therapy Modalities; Occupational Therapy; Capacity Building

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Rehabilitation self-management group, on-line self monitoring of physical function, and organizational capacity building.
  Interventions: Behavioral: Physiotherapy; Behavioral: Occupational Therapy; Behavioral: Capacity Building
- Case matched controls (No Intervention): Usual care in primary health care.

INTERVENTIONS:
Behavioral: Physiotherapy — group self-management classes
  Arms: Intervention Group
Behavioral: Occupational Therapy — group self-management classes
  Arms: Intervention Group
Behavioral: Capacity Building — workshops and case reviews with primary health care team members
  Arms: Intervention Group

SUMMARY:
People who have long-term conditions such as heart disease, diabetes, arthritis etc. face challenges in staying active and able to participate in activities that are important to them. There is some research that suggests that a care model that focuses on physical functioning and helping patients to manage their own conditions will assist them to stay active and healthy longer. In this project, the investigators are testing whether physiotherapy and occupational therapy offered to groups of patients and information about rehabilitation offered to other members of the health care team can help people with chronic conditions to maintain their physical abilities.

DETAILED DESCRIPTION:
Participants older than 44, with at least one chronic disease, (n=60) will participate in a before-and-after study integrating a population based, rehabilitation-focused program targeting physical function into a Family Health Team. The program, delivered by a Physiotherapist and Occupational Therapist, will consist of comprehensive functional assessments and individualized self-management care plans; a rehabilitation based chronic disease self-management program; and on-line self-monitoring of physical function. Process and outcome measures will be administered at baseline and 4 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 44 years and older
* 1 or more chronic conditions
* 3 visits to physician in the past year
* access or willingness to access email

Exclusion Criteria:

* none

Min Age: 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Richardson, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster Family Health Team (Stonechurch Family Health Centre and McMaster Family Practice), Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Richardson J, Letts L, Chan D, Officer A, Wojkowski S, Oliver D, Moore A, McCarthy L, Price D, Kinzie S. Monitoring physical functioning as the sixth vital sign: evaluating patient and practice engagement in chronic illness care in a primary care setting--a quasi-experimental design. BMC Fam Pract. 2012 Apr 3;13:29. doi: 10.1186/1471-2296-13-29. PMID 22471378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two distinct locations of the McMaster Family Health Team.
Period: Overall Study
Arm/Group | Intervention Group | Case Matched Controls
Started | 65 | 59
Completed | 55 | 55
Not Completed | 10 | 4
Not completed — Lost to Follow-up | 6 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Ill health | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Case Matched Controls | Total
Number analyzed (Participants) | 65 | 59 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 37 | 77
  >=65 years | 25 | 22 | 47
Age Continuous [Mean (Standard Deviation); unit: years] | 63.57 (11.81) | 62.62 (10.48) | 63.08 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 85
  Male | 22 | 17 | 39
Region of Enrollment [Number; unit: participants]
  Canada | 65 | 59 | 124

OUTCOME MEASURES:

1. Primary Outcome: Physical Functioning Inventory (PFI)
Description: The PFI is used to assess physical functioning in older adults. It contains 21 tasks from 4 subscales: activities of daily living, instrumental activities of daily living, mobility, moderate activities. A series of questions is used to determine whether the person experiences difficulty in completing a task, the level of difficulty they experience, and any changes to the method and/or frequency of task performance. The PFI is sensitive to steps in the natural history of functional decline that are often not assessed clinically. Range of scores: 0 (most difficulty); 100 (least difficulty).
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Case Matched Controls
Number analyzed (Participants) | 65 | 59
units on a scale | 5.50 (12.14) | 2.96 (10.81)

2. Secondary Outcome: Self-rated Health
Time Frame: 4 months
Reporting Status: Not Posted

3. Secondary Outcome: Health Care Utilization
Time Frame: 4 months
Reporting Status: Not Posted

4. Secondary Outcome: Self-efficacy for Chronic Disease Scale
Time Frame: 4 months
Reporting Status: Not Posted

5. Secondary Outcome: Rapid Assessment of Physical Activity
Time Frame: 4 months
Reporting Status: Not Posted

6. Secondary Outcome: Grip Strength
Time Frame: 4 months
Reporting Status: Not Posted

7. Secondary Outcome: Two Minute Walk Test
Time Frame: 4 months
Reporting Status: Not Posted

8. Secondary Outcome: Patient Assessment of Chronic Illness Care
Time Frame: 4 months
Reporting Status: Not Posted

9. Secondary Outcome: Primary Care Resources and Supports
Time Frame: 4 months
Reporting Status: Not Posted

10. Secondary Outcome: Balance Screen
Time Frame: 4 months
Reporting Status: Not Posted

11. Secondary Outcome: Eight Foot Walk Test
Time Frame: 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intervention Group | Case Matched Controls
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/59
Other Adverse Events (participants affected / at risk) | 0/65 | 0/59

LIMITATIONS AND CAVEATS:
The limited duration of the study period may not allow sufficient time to show the difference in outcome measures such as self-rated health and health care utilization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No